CLINICAL TRIAL: NCT03843892
Title: Expanded Access Use of OFEV (Nintedanib) in Non-IPF Interstitial Lung Disease
Brief Title: An Expanded Access Program to Provide Nintedanib to Patients With Non-IPF ILD Who Have no Alternative Treatment Possibilities
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0380
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: OFEV — twice daily

SUMMARY:
This Expanded Access Program is intended to facilitate the availability of OFEV to patients suffering from non Idiopathic Pulmonary Fibrosis-Interstitial Lung Disease (non IPF-ILD) with a progressive clinical course despite Standard of Care treatment and for whom no satisfactory authorised alternative therapy exists or who cannot enter a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

None

Exclusion Criteria:

- Patients who are eligible for and can participate in an ongoing non Idiopathic Pulmonary Fibrosis-Interstitial Lung Disease (non IPF-ILD) study will be excluded from participation in this Expanded Access Program (EAP).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Banner University Medical Center Tucson, Tucson, Arizona
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - University of Rochester Medical Center, Rochester, New York
  - Centra Medical Group, Bedford, Virginia
  - Inova Fairfax Medical Campus, Falls Church, Virginia